CLINICAL TRIAL: NCT04071756
Title: A Phase II Randomized Double-Blind Trial of Topical Tazarotene 0.1% Gel Versus Placebo Gel for the Prevention of Regorafenib-Induced Hand-Foot-Skin Reaction
Brief Title: Topical Tazarotene Vs Placebo In Hand-Foot-Skin Reactions
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty with patient recruitment
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Nicole LeBoeuf, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19-099
Record Dates: First submitted 2019-06-05; First posted 2019-08-28 (Actual); Results first posted 2023-11-15 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Solid Tumor; Hand-Foot Skin Reaction (HFSR)
Keywords: Solid Tumor; Hand-Foot Skin Reaction (HFSR)
MeSH Terms: interventions — tazarotene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Topical Tazarotene 0.1% Gel Plus BPS (Experimental): * Pharmacy teaching call
  * DFCI approved teaching sheets will be provided
  * 20% urea applied to the palms and soles in the morning + tazarotene 0.1% gel, applied to the palms and soles nightly
  Interventions: Drug: Topical Tazarotene
- Placebo Gel Plus BPS (Placebo Comparator): * A substance that has no therapeutic effect, used as a control in testing new drugs
  * Pharmacy teaching call
  * DFCI approved teaching sheets will be provided
  * 20% urea applied to the palms and soles in the morning with placebo gel applied in the evening.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Topical Tazarotene — This medicine works by making the skin less inflamed and reducing the thickness and pain from lesions of the skin
  Other Names: Tazorac
  Arms: Topical Tazarotene 0.1% Gel Plus BPS
Other: Placebo — A substance that has no therapeutic effect, used as a control in testing new drugs
  Arms: Placebo Gel Plus BPS

SUMMARY:
This research is studying the preventative use of topical 0.1% tazarotene gel daily in addition to best practice standards to reduce the development of hand-foot skin reaction (HFSR).

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The U.S. Food and Drug Administration (FDA) has not approved tazarotene for specifically for hand-foot skin reaction but it has been approved for other uses.

In this research study, the investigators are:

-aiming to determine if the use of tazarotene gel daily, in addition to best practice standards:

* reduces the development of HFSR.
* decreases modification of regorafenib dose due to HFSR
* improves health-related quality of life associated with HFSR
* decreases stress associated with HFSR

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed solid tumors with a plan to initiate regorafenib, or having started regorafenib in the last 48 hours, via dose escalation protocol describe in the ReDOS study in CRC. The ReDOS study recommends this dose escalation of regorafenib:80mg daily x 1 week, 120mg daily x 1 week, 160mg daily times one week, off week, then 160mg daily goal, or maximum tolerated dose thereafter. This is not a separate study; this is the current standard of care for regorafenib dosing. In addition, to compare across the cohorts, patients must be ambulatory with full use of all 4 distal extremities.
* Age ≥ 18
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* Participants must have sufficient organ and marrow function in the opinion of the treating investigator. This can be based on lab reports from an outside facility.
* Women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation Tazarotene is known to be teratogenic, although the dose required with topical application to affect the developing human fetus is unknown. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of administration.
* Women of child-bearing potential (WOCBP) must have a negative serum pregnancy test.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Regorafenib use in combination with another TKI (unless regorafenib was started in the last 48 hours)
* Pregnancy or non-compliance with contraception (4 weeks before, during and for at least 3 ovulatory cycles after treatment cessation). Pregnant women are excluded from this study because tazarotene is category X with the potential for teratogenic or abortifacient effects.
* Nursing or lactating: Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with tazarotene, breastfeeding should be discontinued if the mother is treated.
* A history of hypervitaminosis A
* Other systemic retinoids needed for another condition (ie. Isotretinoin for inflammatory acne, acitretin for psoriasis, bexarotene for CTCL).
* Need for treatment dose systemic steroids or systemic immunosuppressive agents (i.e., for autoimmune disease or cerebral edema) at the time of enrolment
* Psoriasis or other autoimmune disease requiring skin directed or systemic therapy known to impact keratinocyte proliferation (UV therapy to the hands or feet, TNF inhibitors, etc).
* Active skin disease of the hands or feet with redness, scaling or blisters prior to enrolment
* Participants who have had any systemic chemotherapy or immunotherapy within 4 weeks prior to entering the study AND who have not recovered from adverse events on the hands and feet due to the agents administered.
* Participants who are receiving any other investigational agents to treat HFSR.
* Uncontrolled intercurrent illness including, but not limited to, uncontrolled lower extremity edema, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2021-06-12 (Actual); Study Completion 2022-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole LeBoeuf, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BCH - Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email TIDO@childrens.harvard.edu BIDMC - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu MGH - Contact the Partners Innovations team at http://www.partners.org/innovation

RESULTS

PARTICIPANT FLOW:
Groups:
- Topical Tazarotene 0.1% Gel Plus BPS: * Pharmacy teaching call
  * DFCI approved teaching sheets will be provided
  * 20% urea applied to the palms and soles in the morning + tazarotene 0.1% gel, applied to the palms and soles nightly
  Topical Tazarotene: This medicine works by making the skin less inflamed and reducing the thickness and pain from lesions of the skin
- Placebo Gel Plus BPS: * A substance that has no therapeutic effect, used as a control in testing new drugs
  * Pharmacy teaching call
  * DFCI approved teaching sheets will be provided
  * 20% urea applied to the palms and soles in the morning with placebo gel applied in the evening.
  Placebo: A substance that has no therapeutic effect, used as a control in testing new drugs
Period: Overall Study
Arm/Group | Topical Tazarotene 0.1% Gel Plus BPS | Placebo Gel Plus BPS
Started | 5 | 3
Patient Reported Outcomes (PRO) Evaluable | 2 | 1
Completed | 5 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topical Tazarotene 0.1% Gel Plus BPS | Placebo Gel Plus BPS | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (11.1) | 44.0 (18.0) | 55.0 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 3 | 1 | 4
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 8
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 23.3 (3.5) | 30.4 (7.1) | 26 (5.9)

OUTCOME MEASURES:

1. Primary Outcome: Grade 2 or Higher Hand-Foot Skin Reaction (HFSR) Rate
Description: Grade 2 or higher hand-foot skin reaction (HFSR) Rate defined as the percentage of patients in each arm who develop grade-2 or higher HFSR within the first 8 weeks of protocol therapy. Measured via examination by a Dermatology Provider and grading according to CTCAE version 5.
Time Frame: Up to 8 weeks
Measure: Number; unit: percent of participants
Arm/Group | Topical Tazarotene 0.1% Gel Plus BPS | Placebo Gel Plus BPS
Number analyzed (Participants) | 5 | 3
percent of participants | 20 | 33.33

2. Primary Outcome: All Grade Hand-Foot Skin Reaction (HFSR) Rate
Description: Any grade hand-foot skin reaction (HFSR) Rate defined as the percentage of patients in each arm who develop HFSR within the first 8 weeks of protocol therapy. Measured via examination by a Dermatology Provider and grading according to CTCAE version 5.
Time Frame: Up to 8 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Topical Tazarotene 0.1% Gel Plus BPS | Placebo Gel Plus BPS
Number analyzed (Participants) | 5 | 3
percentage of participants | 100 | 100

3. Secondary Outcome: Change in HFS-14 Score From Baseline to Day 56
Description: HFS-14 is a specific quality of life scale developed for patients suffering from Hand-Foot Syndrome. It involves 14 questions per protocol Appendix D. Answers are ranked based on the subscripts listed from the level that affect quality of life much to less. Answers are ranked based on the subscripts from survey to not affect life quality (1-4). Maximum score is 44, and minimum score is 14. Change measured from baseline and day 56. Higher score means worse situation.
Time Frame: At baseline and at day 56.
Population: Trial was terminated at enrollment of 8 participants including n=3 on the placebo arm; the PRO evaluable sample for the placebo arm is not provided due to patient privacy.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Topical Tazarotene 0.1% Gel Plus BPS | Placebo Gel Plus BPS
Number analyzed (Participants) | 2 | 0
units on a scale | 1 [0 to 2] |

4. Secondary Outcome: Change in Perceived Stress Scale (PSS) From Baseline to Day 56
Description: PSS is a classic stress assessment instrument that helping understand how different situations affect patients' feelings and perceived stress. Patients answer 10 questions defined in protocol appendix D. Answers are ranked 0-4. The higher the overall scores indicate higher perceived stress. Score range is from 0 to 40. Higher score means more stressful. Change measured at baseline and day 56.
Time Frame: at baseline and day 56
Population: as for outcome 3
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Topical Tazarotene 0.1% Gel Plus BPS | Placebo Gel Plus BPS
Number analyzed (Participants) | 2 | 0
units on a scale | 7.5 [0 to 13] |

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Of the eight participants enrolled, six reported one or more adverse events (Placebo:2, Tazarotene:4), and two reported no adverse events. All events were classified as either "unrelated" or "unlikely related" to study therapy. In the table below, each participant is classified according to the worst grade reported for each adverse event type. All events were grade 1 or 2.
Arm/Group | Topical Tazarotene 0.1% Gel Plus BPS | Placebo Gel Plus BPS
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/3
Other Adverse Events (participants affected / at risk) | 5/5 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topical Tazarotene 0.1% Gel Plus BPS (N=5) | Placebo Gel Plus BPS (N=3)
Biliary stent blockage (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topical Tazarotene 0.1% Gel Plus BPS (N=5) | Placebo Gel Plus BPS (N=3)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — Grade 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Grade 1
psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — grade 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) — grade 1-2
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — grade 1
rash, maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated prematurely on 7/14/2022 as there had been significant difficulty with patient recruitment.

This report includes data for eight (8) randomized participants. The first enrolled on December 30, 2019, and the last on July 28, 2020.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/56/NCT04071756/Prot_SAP_000.pdf